CLINICAL TRIAL: NCT05700890
Title: Adaptation of the World Health Organization Surgical Safety Checklist to High-Income Healthcare Settings - Phase III: Site Testing Study
Brief Title: The Surgical Safety Checklist Revisited
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ariadne Labs (Other); National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: REB21-0099
Record Dates: First submitted 2022-11-30; First posted 2023-01-26 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Surgical Procedure, Unspecified; Communications Personnel; Tool Use Behavior
Keywords: Surgical Safety Checklist; Patient Safety; Quality improvement; Teamwork; Psychological safety
MeSH Terms: conditions — Communication; Tool Use Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Implementation Team: The Implementation Group will complete two surveys at the beginning of the study, then at five different points during the HPC Toolkit's use, and again three months post-intervention. The surveys are the Safe Surgery Checklist Culture Survey and the SSC Use and Attitudes Survey and a series of user experience surveys.
  They will also do interviews pre- and post-HPC toolkit, and we will observe the Implementation Team's meetings as they work through the toolkit.
- OR Team: The OR members will complete the same pre- and post-intervention surveys (Safe Surgery Checklist Culture Survey and the SSC Use and Attitudes Survey) and do interviews before and after the IT has worked through the HPC toolkit.
- Surgical Patients: Surgical patients will be invited to participate in focus groups on their experiences from the time they enter the hospital on the day of their surgery to the moment they are put under anaesthesia.

SUMMARY:
The goal of this study is to develop and iteratively improve a toolkit - the "High-Performance Checklist" (HPC) toolkit - that provides clinicians with evidence-informed strategies for improving their Modification, Implementation, Training on, and Evaluation of the Surgical Safety Checklist.

The study team will test the toolkit in the operating rooms of Calgary's Peter Lougheed Centre and collect feedback via surveys and questionnaires. This feedback will be used to iteratively improve the toolkit.

By improving clinicians' ability to modify their SSC, the study team hopes to see improvements in its uptake and surgical outcomes for patients.

Participants will be surgical clinical staff members and hospital administration, as well as participants over the age of 18, who have undergone a surgery in the last 90 days. They will all complete the following tasks:

Online or paper questionnaire Semi structured interviews Team meetings

DETAILED DESCRIPTION:
This study is the third phase of a multi-year, multi-stage research project aimed at successful use of the World Health Organization's Safe Surgery Checklist. The study's first stage involved collecting perceptions of the SSC from surgical personnel in five high-income countries: Australia, the United States, Canada, the United Kingdom, and New Zealand. In that stage, interviews and surveys were conducted with individuals who use the SSC. Our results showed barriers and facilitators to the SSC's use and highlighted clinicians' attitudes towards it. The first stage of our study identified the need to better tailor the SSC checklists to meet contextual needs and ongoing gaps in leadership and team performance.

The study's second stage involved building a toolkit aimed at addressing four areas (Modification, Implementation, Training, and Evaluation) through the creation of working groups for each area. These working groups comprised Subject-Matter Experts (SMEs) from the consensus meeting and individuals from the surgical safety field. The output generated by these groups through a consensus-building process is the "High-Performance Checklist" Toolkit ("Toolkit"). The Toolkit is built using the Explore, Prepare, Implement, and Sustain (EPIS) framework and provides clinicians a mechanism for effectively customizing their SSC to their needs.

The third stage of the study involves pilot testing the Toolkit at three different sites and assessing its impact and usefulness in helping implementation teams at these sites. The three sites selected for this study are facilities of different size and scale, for which impact, outcomes, and clinician feedback from Implementation Teams from each site will be compared. The first site is the Peter Lougheed Centre in Calgary, Alberta, then the team intend to run the study at the University of Alberta Hospital and the hospital in Fort McMurray, Alberta.

At each site, three types of participants will be recruited: Implementation team ("ImT") members, operating room ("OR") personnel, and surgical patients. The ImT members will work through the Toolkit to customize their SSC, then the OR personnel will use the modified SSC. The patients will participate in Focus Groups to explore their perceptions of the SSC's use at each site.

From there, we will endeavour to make alterations to the toolkit, if necessary, before rolling it out on a larger scale.

The anticipated result is that clinicians' use of this toolkit will enhance their ability to effectively modify, implement, train, and evaluate their SSC, improve their use of SSC to reduce the rate of adverse events with patients in the OR. It is predicted that the Toolkit will have a positive impact on the culture of patient safety and staff members' perception of psychological safety in the OR.

This study aims to fill the gap in effective checklist modification, training, implementation, and evaluation that was observed during data gathering stage. The study team will gain insight on the utility of a tool designed for improving surgical teams' use of the SSC: how it works, users' perceptions of it, areas for improvement, and ideas for spreading the tool's usage.

Methods: During this stage of the study, the Toolkit will be implemented at the aforementioned Albertan sites. Using an effectiveness-implementation hybrid design, a mixed-methods approach will be applied to assess the implementation of the Toolkit and users' experiences with it. The impact of the toolkit's use on clinical outcomes will also be assessed through the collection of health systems data. Through a series of surveys, interviews, and observations of the toolkit being used, the toolkit's usability, feasibility, and acceptability, and impact on safety culture will be measured before, during, and after the toolkit's implementation. Throughout the study, ratings of the SSC's performance will be taken to assess the toolkit's impact on OR participants' teamwork and SSC engagement.

Operationally, this stage of the study comprises four phases: initial introductions and pre-study data collection, use of the Toolkit by completing the EPIS elements, post-implementation data collection, and a three-months post-implementation follow-up. Data will be collected during each phase to assess the impact of the toolkit and the experience of its users.

Data analysis: survey, health systems data, and SSC performance ratings will be analyzed using SPSS and qualitative data from the observations and interviews will be analyzed thematically using NVIVO.

ELIGIBILITY:
Inclusion Criteria:

* surgeons, anesthesiologists, nurses and administrator will be included in the study
* surgical patients that have undergone surgery within the last three months at the Peter Lougheed Centre

Exclusion Criteria:

* Patients that are unable to fill out a survey or participate in a semi structured interview
* Patients that surgery was done more than 3 months ago
* Surgical patients that are under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are three types of participants in this study:
  1. The Implementation Team includes physicians, nurses, administrators, and patient advocates
  2. The OR Team
  3. Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Perception of the HPC Toolkit | the initial 8 weeks of interacting with the study site
  We will assess if the clinicians use of the HPC toolkit foster improvement in their use of the SSC. Surveys and semi-structured interviews will be collected at baseline, after the HPC introduction and at follow-up to assess if the HPC toolkit is sustained.
Reduction rate of adverse events in patient | Through study completion, and average of 1 year
  We will assess if the clinicians use of the HPC toolkit reduces the rate of adverse events in patients
SSC Attitudes and OR Culture | Approximately the first and last 8 weeks interacting with the study site.
  The Implementation Team ("ImT") and OR Team's perceptions of the SSC and OR Culture will be measured through surveys at3 points in time.
Patient Surgical Experiences Survey | Approximately the first and last 8 weeks interacting with the study site.
  Patients' experiences with surgery before and after the HPC Toolkit's implementation.
User Experience Surveys | Approximately the first and last 8 weeks interacting with the study site
  The ImT's experiences with the HPC Toolkit: ease of use, intuitiveness, layout, etc.
CheckPOINT observation tool | Approximately the first and last 8 weeks interacting with the study site
  In situ observations of the SSC's use in the OR; measures SSC use in practice. Captured by the ImT and OR Team participants.
Semi-structured interviews | Approximately the first and last 8 weeks interacting with the study site
  Participants' perceptions of the SSC and the HPC Toolkit's impact on it
Meeting observations | up to 16 weeks
  The Implementation Team's use of the HPC Toolkit

SECONDARY OUTCOMES:
Healthcare system data collection | Up to 2 years
  AHS data analytics will be collected to assess the HPC toolkit's impact on patient safety and clinical throughput.
Measures of surgical safety | Up to 2 years
  Health systems data will be collected to look at the following perioperative events:a. Surgical Site Infection Rate (%) b. 30-Day In Hospital Mortality after major surgery (crude and risk adjusted) c. 30-Day re-admission after surgery (crude rate and risk adjusted rate) d. Unplanned ED visit within 30 days after surgery (%) e. Unplanned Re-Operative events (%) - within 24 hours? f. Peri-operative venous thromboembolism (VTE) diagnosis (%)
Effectiveness of SSC practice | Up to 2 years
  Errors averted by using the safe Surgery Checklist (Provincial Data):a. Site/Side/Location/Procedure - Incomplete or incorrect b. Pre op prep/lab/meds - incomplete or incorrect c. Equipment/Supplies - Missing or incorrect d. Allergies/Contraindications - to medication/equipment e. Documentation/history - incomplete or incorrect f. Wrong patient g. Not specified These data will be collected before and after implementation of the High Performance Toolkit to demonstrate the effectiveness of SSC practice.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Brindle, MD, Principal Investigator — University of Calgary
Locations (1):
- Karolina Kogut, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Background] Campbell S, Greenwood M, Prior S, Shearer T, Walkem K, Young S, Bywaters D, Walker K. Purposive sampling: complex or simple? Research case examples. J Res Nurs. 2020 Dec;25(8):652-661. doi: 10.1177/1744987120927206. Epub 2020 Jun 18. PMID 34394687
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Delisle M, Pradarelli JC, Panda N, Koritsanszky L, Sonnay Y, Lipsitz S, Pearse R, Harrison EM, Biccard B, Weiser TG, Haynes AB; Surgical Outcomes Study Groups and GlobalSurg Collaborative. Variation in global uptake of the Surgical Safety Checklist. Br J Surg. 2020 Jan;107(2):e151-e160. doi: 10.1002/bjs.11321. PMID 31903586
- [Background] Devcich DA, Weller J, Mitchell SJ, McLaughlin S, Barker L, Rudolph JW, Raemer DB, Zammert M, Singer SJ, Torrie J, Frampton CM, Merry AF. A behaviourally anchored rating scale for evaluating the use of the WHO surgical safety checklist: development and initial evaluation of the WHOBARS. BMJ Qual Saf. 2016 Oct;25(10):778-86. doi: 10.1136/bmjqs-2015-004448. Epub 2015 Nov 20. PMID 26590200
- [Background] Dixon E, Vollmer CM Jr, Bathe O, Sutherland F. Training, practice, and referral patterns in hepatobiliary and pancreatic surgery: survey of general surgeons. J Gastrointest Surg. 2005 Jan;9(1):109-14. doi: 10.1016/j.gassur.2004.03.008. PMID 15623451
- [Background] Fourcade A, Blache JL, Grenier C, Bourgain JL, Minvielle E. Barriers to staff adoption of a surgical safety checklist. BMJ Qual Saf. 2012 Mar;21(3):191-7. doi: 10.1136/bmjqs-2011-000094. Epub 2011 Nov 7. PMID 22069112
- [Background] Halcomb EJ, Davidson PM. Is verbatim transcription of interview data always necessary? Appl Nurs Res. 2006 Feb;19(1):38-42. doi: 10.1016/j.apnr.2005.06.001. PMID 16455440
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Dziekan G, Herbosa T, Kibatala PL, Lapitan MC, Merry AF, Reznick RK, Taylor B, Vats A, Gawande AA; Safe Surgery Saves Lives Study Group. Changes in safety attitude and relationship to decreased postoperative morbidity and mortality following implementation of a checklist-based surgical safety intervention. BMJ Qual Saf. 2011 Jan;20(1):102-7. doi: 10.1136/bmjqs.2009.040022. PMID 21228082
- [Background] King DK, Shoup JA, Raebel MA, Anderson CB, Wagner NM, Ritzwoller DP, Bender BG. Planning for Implementation Success Using RE-AIM and CFIR Frameworks: A Qualitative Study. Front Public Health. 2020 Mar 3;8:59. doi: 10.3389/fpubh.2020.00059. eCollection 2020. PMID 32195217
- [Background] Laugaland K, Aase K, Waring J. Hospital discharge of the elderly--an observational case study of functions, variability and performance-shaping factors. BMC Health Serv Res. 2014 Aug 30;14:365. doi: 10.1186/1472-6963-14-365. PMID 25175924
- [Background] Lepanluoma M, Takala R, Kotkansalo A, Rahi M, Ikonen TS. Surgical safety checklist is associated with improved operating room safety culture, reduced wound complications, and unplanned readmissions in a pilot study in neurosurgery. Scand J Surg. 2014 Mar;103(1):66-72. doi: 10.1177/1457496913482255. Epub 2013 Dec 17. PMID 24345978
- [Background] Moullin JC, Dickson KS, Stadnick NA, Rabin B, Aarons GA. Systematic review of the Exploration, Preparation, Implementation, Sustainment (EPIS) framework. Implement Sci. 2019 Jan 5;14(1):1. doi: 10.1186/s13012-018-0842-6. PMID 30611302
- [Background] Russ SJ, Sevdalis N, Moorthy K, Mayer EK, Rout S, Caris J, Mansell J, Davies R, Vincent C, Darzi A. A qualitative evaluation of the barriers and facilitators toward implementation of the WHO surgical safety checklist across hospitals in England: lessons from the "Surgical Checklist Implementation Project". Ann Surg. 2015 Jan;261(1):81-91. doi: 10.1097/SLA.0000000000000793. PMID 25072435
- [Background] Solsky I, Berry W, Edmondson L, Lagoo J, Baugh J, Blair A, Singer S, Haynes AB. World Health Organization Surgical Safety Checklist Modification: Do Changes Emphasize Communication and Teamwork? J Surg Res. 2020 Feb;246:614-622. doi: 10.1016/j.jss.2018.09.035. Epub 2018 Oct 24. PMID 30528925
- [Background] Stelfox HT, Crimi C, Berra L, Noto A, Schmidt U, Bigatello LM, Hess D. Determinants of tracheostomy decannulation: an international survey. Crit Care. 2008;12(1):R26. doi: 10.1186/cc6802. Epub 2008 Feb 26. PMID 18302759
- [Background] Taylor MJ, McNicholas C, Nicolay C, Darzi A, Bell D, Reed JE. Systematic review of the application of the plan-do-study-act method to improve quality in healthcare. BMJ Qual Saf. 2014 Apr;23(4):290-8. doi: 10.1136/bmjqs-2013-001862. Epub 2013 Sep 11. PMID 24025320
- [Background] Urbach DR, Govindarajan A, Saskin R, Wilton AS, Baxter NN. Introduction of surgical safety checklists in Ontario, Canada. N Engl J Med. 2014 Mar 13;370(11):1029-38. doi: 10.1056/NEJMsa1308261. PMID 24620866
- [Background] Wang Y, Eldridge N, Metersky ML, Verzier NR, Meehan TP, Pandolfi MM, Foody JM, Ho SY, Galusha D, Kliman RE, Sonnenfeld N, Krumholz HM, Battles J. National trends in patient safety for four common conditions, 2005-2011. N Engl J Med. 2014 Jan 23;370(4):341-51. doi: 10.1056/NEJMsa1300991. PMID 24450892
- [Background] AHRQ (2022). "What is Patient Safety Culture?". Agency for Healthcare Research and Quality. Accessed on August 25, 2022.
- [Background] AHS (2021). "Safe Surgery Checklist: Surgery SCN". Alberta Health Services. Accessed on December 21, 2021.
- [Background] DeWalt, K. M., & DeWalt, Billie R. (2011). Participant observation a guide for fieldworkers. Lanham, Md.: Rowman & Littlefield.
- [Background] Laugwitz, B., Held, T, & Schrepp, M. (2008). Construction and Evaluation of a User Experience Questionnaire. USAB 2008. 5298. 63-76. 10.1007/978-3-540-89350-9_6.
- [Background] Lund, A. (2001). Measuring Usability with the USE Questionnaire. Usability and User Experience Newsletter of the STC Usability SIG. 8
- [Background] Miles, M. B., & Huberman, A. M. (1994). Qualitative data analysis: an expanded sourcebook. Thousand Oaks, Calif.: Sage.
- [Background] Minge, M., Thuering, M., Wagner, I., & Kuhr, C. (2017). The meCUE Questionnaire: A Modular Tool for Measuring User Experience. 486. 115-128. 10.1007/978-3-319-41685-4_11.
- [Background] Touchette, A. (2020, May 21). "The Consolidated Framework for Implementation Research (CFIR)". CHI KT Platform. Accessed on February 17, 2022.
- [Background] Urban D, Burian BK, Patel K, Turley NW, Elam M, MacRobie AG, Merry AF, Kumar M, Hannenberg A, Haynes AB, Brindle ME. Surgical Teams' Attitudes About Surgical Safety and the Surgical Safety Checklist at 10 Years: A Multinational Survey. Ann Surg Open. 2021 Jul 6;2(3):e075. doi: 10.1097/AS9.0000000000000075. eCollection 2021 Sep. PMID 36590849
- [Result] Arber A. "Pain talk" in hospice and palliative care team meetings: an ethnography. Int J Nurs Stud. 2007 Aug;44(6):916-26. doi: 10.1016/j.ijnurstu.2006.04.002. Epub 2006 Jun 9. PMID 16764880